CLINICAL TRIAL: NCT04921605
Title: A Clinical Study of Management of Severe Tricuspid Regurgitation With Transcatheter Mitral Valve Clamping System
Brief Title: Feasibility Study of Dragonfly System for Severe Tricuspid Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFly-T-I
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-06

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tricuspid regurgitation (Experimental): Subjects received the Dragonfly system for the treatment of tricuspid regurgitation.
  Interventions: Device: DragonFly transcatheter mitral valve clamping system

INTERVENTIONS:
Device: DragonFly transcatheter mitral valve clamping system — To conduct edge-to-edge repair with Dragonfly System under the guidance of transesophageal echocardiography.

SUMMARY:
The study is designed to assess the feasibility of the DragonFly transcatheter mitral valve clamping system for the treatment of symptomatic severe tricuspid regurgitation.

DETAILED DESCRIPTION:
This study is a prospective, single-center design. Patients are clinically symptomatic patients with severe tricuspid regurgitation despite medical therapy with an expected moderate or greater surgical risk and prohibited to thoracotomy. After signing an informed consent form, subjects are enrolled and treated with the DragonFly Transcatheter Mitral Valve Repair System. All subjects receive clinical follow-up immediately after the procedure, before discharge, and 30 days, 6 months, 12 months and 24 months after the procedure.

Incidence of MAEs at 30 days and immediate procedural success is used as the primary endpoint. The MAEs include device- or procedure-related death, myocardial infarction, stroke, renal failure, and nonelective cardiovascular surgery associated with adverse events. The immediate procedural success is defined as successful implantation of a tricuspid valve-clamp device with at least a one-grade reduction in severity of tricuspid regurgitation at discharge (30-day echocardiography if discharge records were not available or were uninterpretable). Subjects who died or underwent tricuspid valve surgery prior to discharge were defined as immediate procedure failure.

The secondary endpoints include all-cause mortality, cardiovascular-related mortality, the incidence of serious adverse events, heart failure rehospitalization, changes of NYHA classification, reduction of tricuspid regurgitation severity, the proportion of reoperations, changes of quality of life as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) score.

The study comprises two main objectives, firstly, to assess the safety and effectiveness of the DragonFly transcatheter mitral valve clamping system for the treatment of symptomatic severe tricuspid regurgitation despite medical therapy with an expected moderate or greater surgical risk and prohibited to thoracotomy. Secondly, to evaluate the feasibility and performance of the device and to familiarize clinicians with the device and procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subject is medically treated, remains symptomatic and has severe tricuspid regurgitation confirmed by echocardiogram.
3. New York Heart Function Class (NYHA) II-IVa, or hospitalization for heart failure due to one or more episodes in the past 12 months.
4. Patient eligible for transcatheter tricuspid repair as well as suitable for use of the study device.
5. Subject had an expected moderate or greater surgical risk confirmed by the cardiac surgeon, or the subject as not suitable for surgical thoracotomy confirmed by local doctor.
6. Life expectancy ≥ 12 months.
7. Subjects have been informed of the nature of the study, understand the purpose of the clinical trial, voluntarily participate, agree to its provisions, and have provided written informed consent approved by the Ethics Committee.

Exclusion Criteria:

1. Tricuspid valve anatomy not suitable for device positioning or implantation as assessed by the clinical team, including but not limited to the following: a) calcification in the leaflet capture area; b) tricuspid valve perforation defect>2 cm; c) severe tricuspid valve leaflet perforation, fissure and other lesions that preclude device implantation; d) Ebstein malformation.
2. Presence of other serious valvular heart disease requiring intervention such as combined severe aortic stenosis or regurgitation, severe mitral regurgitation. Note: If combined with mitral and tricuspid valve lesions, mitral valve surgery can be selected first, and trial evaluation can be conducted after waiting for 60 days.
3. Tricuspid stenosis, defined as tricuspid valve orifice area ≤ 1.0 cm2 and/or trans-tricuspid pressure difference ≥ 5 mmHg.
4. After tricuspid surgery or tricuspid transcatheter treatment.
5. Echocardiogram suggesting an intracardiac thrombus, vegetation, or mass; implant or thrombus in the femoral vein or inferior vena cava.
6. Left ventricular ejection fraction (LVEF) ≤ 20%.
7. Refractory heart failure requiring advanced intervention (eg, left ventricular assist device, heart transplant) (ACC/AHA stage D heart failure).
8. Pulmonary artery systolic pressure>70 mmHg, or irreversible pre-capillary pulmonary hypertension (measured by right heart catheter).
9. Severe and uncontrolled hypertension: systolic blood pressure (SBP) ≥ 180 mmHg and diastolic blood pressure (DBP) ≥ 110 mmHg.
10. Active endocarditis, active rheumatic heart disease, or rheumatic valvular heart disease leading to tricuspid valve leaflet lesions (poor leaflet compliance, perforation, etc.).
11. After a pacemaker or ICD implantation.
12. Myocardial infarction or unstable angina within 4 weeks; untreated severe coronary stenosis requiring revascularization.
13. Percutaneous coronary intervention was performed within 30 days before surgery.
14. Hemodynamic instability, defined as systolic blood pressure<90mmHg with or without cardiogenic shock or requiring intra-aortic balloon counterpulsation or other hemodynamic support device.
15. Cerebrovascular accident (CVA) within the previous 90 days.
16. Renal failure, currently requiring dialysis.
17. Bleeding disorder or hypercoagulability.
18. Acute peptic ulcer or gastrointestinal bleeding within 3 months prior to surgery.
19. Concurrent treatment contraindication or allergic reaction to dual antiplatelet and anticoagulant drugs. Note: Antiplatelet drugs alone or anticoagulant drugs are contraindicated and not used as exclusion criteria.
20. Active infection, currently requiring antibiotic therapy.
21. Severe chronic obstructive pulmonary disease requiring continuous oxygen inhalation.
22. Known hypersensitivity to device materials.
23. Life expectancy less than 12 months.
24. Pregnant and lactating women, women who are ready to conceive.
25. Patients who have participated in any drug and/or medical device clinical trial within 1 month prior to this trial.
26. Subjects deemed unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | 30days
  Major adverse events included device- or procedure-related death, myocardial infarction, stroke, renal failure, and nonelective cardiovascular surgery associated with adverse events.
Immediate procedural success | up to 30 days
  Defined as successful implantation of a tricuspid valve-clamp device with at least a one-grade reduction in severity of tricuspid regurgitation at discharge (30-day echocardiography if discharge records were not available or were uninterpretable). Subjects who died or underwent tricuspid valve surgery prior to discharge were defined as immediate procedure failure.

SECONDARY OUTCOMES:
All-cause mortality | 12, 24 months
  All-cause mortality included cardiac, non-cardiac, and unexplained death
Cardiovascular-related mortality | 12, 24 months
  Incidence of cardiovascular-related mortality
Serious adverse events | 12, 24 months
  Incidence of serious adverse events
Heart failure rehospitalization | 12, 24 months
  Incidence of heart failure rehospitalization
NYHA classification | 30 days, 6 months, 12 months and 24 months
  Changes of NYHA classification from baseline
Tricuspid regurgitation reduction | 30 days, 6 months, 12 months and 24 months
  Proportion of postoperative reduction in severity of tricuspid regurgitation
Reoperations of Tricuspid regurgitation | 30 days, 6 months, 12 months and 24 months
  Proportion of reoperations for tricuspid regurgitation after procedure
Quality of life assessment | 12, 24 months
  Changes in quality of life as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) score from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD, PH.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No